CLINICAL TRIAL: NCT00142753
Title: Correlates of HBV-Specific B Cell Memory Following Vaccination in HIV-Infected Adolescents and HIV-Uninfected Adolescents: A Substudy of ATN 024 and ATN 025
Brief Title: Immunologic Memory (Supp. of ATN 024)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 048
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: Hepatitis B vaccines; HIV-infected adolescents; Hepatitis B infection
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Engerix-B; twinrix; Recombivax HB

ARMS (5):
- A1: ATN 024 Energix-B Standard Adult Dose (Active Comparator)
  Interventions: Biological: Engerix B
- A2: ATN 024 Engerix-B Increased Adult Dose (Experimental)
  Interventions: Biological: Engerix B
- A3: ATN 024 Twinrix Standard Adult Dose (Active Comparator)
  Interventions: Biological: Twinrix for ATN 024
- B1: ATN 025 Recombivax (Experimental)
  Interventions: Biological: Recombivax
- B2: ATN 025 Twinrix (Experimental)
  Interventions: Biological: Twinrix for ATN 025

INTERVENTIONS:
Biological: Engerix B — Standard adult dose for A1; increased adult dose for A2. Doses at Entry, Weeks 4 and 24. Non-responders (<10 IU/mL of antibody at week 28/4 weeks after dose #3) will receive Engerix-B increased adult dose at Week 48.
  Other Names: There are no other names.
  Arms: A1: ATN 024 Energix-B Standard Adult Dose; A2: ATN 024 Engerix-B Increased Adult Dose
Biological: Twinrix for ATN 024 — Standard adult dosage, taken at Entry, Weeks 4 and 24. Non-responders (<10 IU/mL of antibody at week 28/4 weeks after dose #3) will receive Engerix-B increased adult dose at week 48.
  Other Names: There are no other names.
  Arms: A3: ATN 024 Twinrix Standard Adult Dose
Biological: Recombivax — Dosage at entry and week 24; non-responders ((<10 IU/mL of antibody at week 28/4 weeks after dose #3) will receive 3rd dose of Recombivax during weeks 48-72.
  Other Names: There are no other names.
  Arms: B1: ATN 025 Recombivax
Biological: Twinrix for ATN 025 — Doses at Entry and Week 24. Non-responders (<10 IU/mL of antibody at week 28/4 weeks after dose #3) will receive a dose of Recombivax during week 48-72.
  Other Names: There are no other names.
  Arms: B2: ATN 025 Twinrix

SUMMARY:
This is an exploratory, laboratory-based evaluation of cellular immune response to immunization with hepatitis B surface antigen in HIV-infected and HIV-uninfected adolescents. This is a substudy of ATN 024 and ATN 025. This substudy will compare cellular immune response in responders and nonresponders to immunization and also evaluate the relationship of these factors to the persistence of known correlates of serologic protection for the hepatitis B virus.

DETAILED DESCRIPTION:
This substudy will enroll volunteers from participants of ATN 024 and ATN 025. Participants in ATN 024 are HIV-infected youths aged 12-24 years while participants in ATN 025 are HIV-uninfected youths aged 12-17 years. These youths must also be negative for HBV core antibody, HBV surface antigen, and HBV surface antibody to be eligible.

Blood will be drawn from study participants prior to immunization, 1 month after completion of primary immunization and at study exit (week 72 for ATN 024 and week 76 for ATN 025) for cytokine assays and enumeration of antibody-secreting cells. In addition, the antibody to HBV surface antigen will be determined 2 and 4 weeks after supplemental immunization in nonresponders to the primary series and at study exit.

This laboratory substudy is designed to evaluate some aspects of cellular immune response to hepatitis B vaccination that are directly related to the generation and durability of antibody response to HBV surface antigen in HIV-infected and HIV-uninfected adolescents. Cytokine production by peripheral mononuclear cells will be determined following in-vitro stimulation, and antibody-secreting cells will be enumerated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are eligible for participation in ATN 024 and ATN 025 are eligible for ATN 048. Subjects consented for ATN 024 or ATN 025 should be consented for ATN 048 at the same time. A written informed assent/consent must be obtained from the subject along with written parental/legal guardian permission as determined by the local IRB before any study-related procedures are performed.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To measure interferon-γ (IFN-γ), interleukin -4 (IL-4), and interleukin-10 (IL-10) production in serologic responders and non-responders. | Before and one month after receipt of primary series of immunization.
To measure concentration of hepatitis B antibodies in serologic responders and non-responders. | 1, 2, and 4 weeks after supplemental vaccine dose.
To measure concentration of antibody-secreting cells in serologic responders and non-responders. | Before and one month after receipt of primary series of immunization.

SECONDARY OUTCOMES:
Measure whether the profile of cytokine secretion or the number of antibody-secreting cells can be used as a predictor of anamnestic response to a supplemental vaccine dose following serologic nonresponse to a primary series of immunization. | Prior to immunization, 1 month after primary immunization, at study exit (week 72 for ATN 024; week 76 for ATN 025); at 2 & 4 weeks after supplemental immunization in nonresponders, & at study exit for ATN 024 subjects.
To compare the rate of loss of antibody-secreting cells after vaccination through the end of the study in each vaccine arm. | Prior to immunization, 1 month after completion of primary immunization and at study exit.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Obaro, MBBS, PhD, Study Chair — ATN
Locations (4):
- United States (4):
  - Childrens Hosp of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Franciso, California
  - Children's Hosp Natinal Med Center, Washington D.C., District of Columbia
  - Tulane Med Center, New Orleans, Louisiana

REFERENCES:
- See also: (Website for the Adolescent Trials Network for HIV/AIDS Interventions) — http://www.atnonline.org